CLINICAL TRIAL: NCT01054391
Title: NEC Trial - Nfocus - Neurovascular Embolization Cover for Treatment of Intracranial Aneurysms and Carotid/Vertebrobasilar Fistulae - A Non-Randomized Pilot Study
Brief Title: Neurovascular Embolization Cover for Treatment of Intracranial Aneurysms and Carotid/Vertebrobasilar Fistulae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nfocus Neuromedical (Industry)
Responsible Party: Tom Ross, Vice-President, Nfocus Neuromedical Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEC001
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Intracranial Aneurysms; Cavernous Carotid Fistula; Vertebrobasilar Fistula
MeSH Terms: conditions — Intracranial Aneurysm; Carotid-Cavernous Sinus Fistula

ARMS (1):
- NEC Arm (Experimental): Utilization of NEC (Neurovascular Embolization Cover) for the treatment of intracranial aneurysms and carotid/vertebrobasilar fistulae
  Interventions: Device: NEC - Neurovascular Embolization Cover

INTERVENTIONS:
Device: NEC - Neurovascular Embolization Cover — Implantation of NEC for the treatment of intracranial aneurysms and carotid/vertebrobasilar fistuale arising from a parent vessel of 2.5 to 4.5mm

SUMMARY:
The purpose of this study is to determine whether the NEC device can effectively occlude the intracranial aneurysm or the carotid/vertebrobasilar fistula and maintain parent vessel patency

DETAILED DESCRIPTION:
SAH (subarachnoid hemorrhage) is a devastating medical emergency. As many as 60% of patients who are afflicted die in the first 30 days as a result of the SAH, or remain severely disabled from the bleed. Existing treatment options include: medical management; endovascular therapy and surgical therapy. Endovascular techniques using detachable coils have now been refined to include stents which serve to prevent the coil mass from dislodging. Further improvement is believed to be possible with the NEC which creates a seal to exclude the aneurismal lumen from blood flow without the need for coils. This study involves the endovascular placement of the NEC across the aneurysm neck in order to treat a subset of aneurysms without coils.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unruptured aneurysm OR ruptured aneurysm in clinically stable patients in whom coils alone are not an efficient treatment in the opinion of the investigator (i.e., large neck or fusiform aneurysm) OR direct fistulae (Type A - traumatic or aneurismal) and indirect if dural branches come from the internal carotid or vertebral artery and cannot be embolized selectively
* Subject has a confirmed diagnosis of an intracranial (including intracavernous and intrapetrous regions) sidewall saccular aneurysm or carotid vertebrobasilar fistula
* Parent artery reference diameter is >2.5mm and <4.5mm
* Subject is an adult above age 18
* Subject is able to provide written Informed Consent
* Subject has good general health, is clinically stable, and is considered to be mentally sound
* Subject is able and is willing to meet all expected requirements of the clinical protocol, including attending the scheduled follow-up examinations for the duration of this trial.

Exclusion Criteria:

* Subject has subarachnoid hemorrhage (SAH) < three (3) weeks prior to NEC procedure
* Subject has had prior stenting of the target aneurysm.
* Subject is contraindicated for antiplatelet therapy,anticoagulant therapy, or radiographic contrast media.
* Subject has collagen vascular disease.
* Subject has a contraindication to angiography (e.g., serum creatinine level > 2.5 mg/dL)
* Subject has evidence of active infection at the time of treatment
* Subject is pregnant or breastfeeding or unwilling to use birth control for duration of study
* Subject has participated in a study involving an investigational drug or device within 30 days prior to proposed entry into subject study
* Subject is unable to comply with study procedures or protocol
* Subject has co-morbid disease or condition expected to compromise survival or ability to complete follow-up assessments to 180 days

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who show complete occlusion of target aneurysm or or fistula as judged by Core Laboratory radiologist by angiography | 6 month follow-up
Proportion of subjects who experience neurologic death or ipsilateral stroke | 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Olav Jansen, Prof. Dr. med., Principal Investigator — Universitatsklinikum Schleswig-Holstein Campus Kiel Institut fur Neuroradiologie
Locations (2):
- Germany (2):
  - Universitatsklinikum Schleswig-Holstein Campus Kiel Institut fur Neuroradiologie, Kiel
  - Universitatsklinikum Schleswig-Holstein Institut fur Neuroradiologie, Lübeck